CLINICAL TRIAL: NCT00155727
Title: Comparison of Treatment Outcome for Laparoscopic Colectomy Versus Traditional Open Colectomy for the Treatment of Colorectal Cancer: … A Prospective Randomized Clinical Trial
Brief Title: Comparison of Laparoscopic Colectomy Versus Open Colectomy for Colorectal Cancer: … A Prospective Randomized Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9100017028
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2005-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer, laparoscopic colectomy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The laparoscopic colectomy has been enthusiastically used by many colorectal surgeons in Taiwan, Japan, Europe, and USA, for around 10 years. Further clarification of the controversies cited above will be based on the evidence-based medicine, i.e., the randomized, well-controlled, prospective clinical trials. Actually, a handful of randomized prospective data regarding the laparoscopic colectomy has been appeared in USA and Europe. However, we still do not have this kind of data in Taiwan, and therefore this study is important and mandatory.

In this project, we assumed that a difference in cancer-related survival of less then 15% between treatments indicates an equivalent efficacy. Assuming a 70% 5-year, cancer-related survival of stage II and III colorectal cancer patients in the open colectomy group, a minimum of 100 patients per group was required to showed that both surgical techniques were equivalent with an α-level of 0.20 and a β error of 0.05. Only patients with stage II and III disease undergoing curative resection will be enrolled onto this study. The patients will be randomly allocated to either treatment group by block randomization method. Postoperatively, the patients will be prospectively evaluated regarding the following parameters including operative stress, such as erythrocyte sedimentation rate, serum interleukin-6, WBC counts and classification, CD-4 to CD-8 ratio, postoperative life quality, such as wound size, degree of pain, time to have flatus passage and feeding, time to resume daily activity and work, and the oncological outcomes, such as recurrence patterns of tumor, and 5-year patient survival. The evaluation of above-mentioned parameters will be single-blindly done by our research assistant, who has no idea of both surgical techniques. We hope this study will promote the level of surgical research in Taiwan.

DETAILED DESCRIPTION:
The appropriateness of laparoscopic surgery for the resection of colorectal cancer has been the focus of controversy. The pros insist that besides the smaller wound size, laparoscopic colectomy should induce lesser perioperative stress, which was evidenced by the less pain, quicker flatus passage, early feeding, and more rapid to resume daily activity and work. Moreover, since the laparoscopic colectomy induces lesser immunosuppression, this may be potentially positive for the treatment of colorectal cancer patients. However, the cons insist that first of all, when the summation of 4 or 5 ports, and incisional wound to retrieve specimen in laparoscopic colectomy were considered, the total wound size in laparoscopic colectomy is basically similar to that of the open colectomy. Secondly, since the laparoscopic surgeons advocated that the extent of intra-abdominal dissection was the same between laparoscopic and open colectomy, it seems illogical to speculate that laparoscopic procedure is less invasive for the colorectal cancer patients than the open procedure. Moreover, in regard of the short-term improvement of life quality (based on the evaluation of parameters including less painful, quicker to have flatus passage, feeding, to resume daily activity, to return to work, etc.), there is no denying that these potential benefits are at the sacrifice of spending more money, and therefore, it is still unknown if laparoscopic colectomy is cost-effective. Thirdly and most important of all, laparoscopic colectomy is a more difficult for most surgeons, and therefore the learning curve is more difficult to overcome. Moreover, many surgeons concerned if pneumoperitoneum during the laparoscopic procedure will reinforce the intraperitoneal spread of colorectal cancer. Based on above-mentioned reasons, many colorectal surgeons hesisted between the lines of safety and efficacy of laparoscopic colectomy.

However, apparently, the laparoscopic colectomy has been enthusiastically used by many colorectal surgeons in Taiwan, Japan, Europe, and USA, for around 10 years. Further clarification of the controversies cited above will be based on the evidence-based medicine, i.e., the randomized, well-controlled, prospective clinical trials. Actually, a handful of randomized prospective data regarding the laparoscopic colectomy has been appeared in USA and Europe. However, we still do not have this kind of data in Taiwan, and therefore this study is important and mandatory.

In this project, we assumed that a difference in cancer-related survival of less then 15% between treatments indicates an equivalent efficacy. Assuming a 70% 5-year, cancer-related survival of stage II and III colorectal cancer patients in the open colectomy group, a minimum of 100 patients per group was required to showed that both surgical techniques were equivalent with an α-level of 0.20 and a β error of 0.05. Only patients with stage II and III disease undergoing curative resection will be enrolled onto this study. The patients will be randomly allocated to either treatment group by block randomization method. Postoperatively, the patients will be prospectively evaluated regarding the following parameters including operative stress, such as erythrocyte sedimentation rate, serum interleukin-6, WBC counts and classification, CD-4 to CD-8 ratio, postoperative life quality, such as wound size, degree of pain, time to have flatus passage and feeding, time to resume daily activity and work, and the oncological outcomes, such as recurrence patterns of tumor, and 5-year patient survival. The evaluation of above-mentioned parameters will be single-blindly done by our research assistant, who has no idea of both surgical techniques. We hope this study will promote the level of surgical research in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted to our unit since January 2000 with adenocarcinoma of the colon and rectum will be assessed.

Exclusion Criteria:

* Cancer with distant metastasis, adjacent organ invasion, intestinal obstruction, past colonic surgery, and no consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2000-01; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung Liang, M.D., Ph.D., Principal Investigator — Department of Surgery, National Taiwan University Hospital, No.7, Chung-Shan South Road, Taipei, TAIWAN, R.O.C.
Locations (1):
- Department of Surgery, National Taiwan University Hospital, No.7, Chung-Shan South Road, Taipei, TAIWAN, R.O.C., Taipei, Taiwan